CLINICAL TRIAL: NCT07117487
Title: A Phase 3 Open-label Study to Evaluate Safety, Tolerability, and Immunogenicity of Revaccination With mRNA-1345 at Least 12 Months Following a Primary Dose of a Licensed Protein Subunit RSV Vaccine in Adult Participants ≥60 Years of Age
Brief Title: A Study of mRNA-1345 Following a Primary Dose of a Licensed Protein Subunit Respiratory Syncytial Virus (RSV) Vaccine in Adult Participants ≥60 Years of Age
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1345-P306
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; Safety; Vaccines
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-1345 (Experimental): Participants will receive a single dose of mRNA-1345 injection administered intramuscularly on Day 1.
  Interventions: Biological: mRNA-1345

INTERVENTIONS:
Biological: mRNA-1345 — Suspension for injection

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and immunogenicity of mRNA-1345 in participants who have been previously vaccinated with either Arexvy or Abrysvo at least 12 months prior to enrollment, are medically stable and aged ≥60 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants may have one or more chronic medical diagnoses, but should be medically stable as assessed by:

  * Absence of changes in medical therapy within 60 days of Visit 1 due to treatment failure or toxicity.
  * Absence of serious or significant medical events within 30 days of Visit 1.
  * Absence of known, current, and life-limiting diagnoses which, in the opinion of the Investigator, would make completion of the protocol unlikely.
* Participant has received a single dose of Arexvy or Abrysvo at least 12 months prior to Visit 1. Participants must provide proof of RSV vaccination status (including brand and date received) prior to enrollment.

Key Exclusion Criteria:

* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤14 days prior to study injection (Day 1) or plans to receive a vaccine authorized or approved by a local health agency within 14 days after the study injection. Nonstudy vaccination(s) should not be delayed.
* Prior participation in research involving receipt of any investigational RSV product (drug/biologic).
* Has received systemic immunoglobulins, long-acting biological therapies that affect immune responses (for example, infliximab) or blood products within 90 days prior to Visit 1 or plans to receive them during the study.

Other protocol-specified inclusion and/or exclusion criteria may apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 up to Day 7 (7 days post-injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Day 1 up to Day 28 (28 days post-injection)
Number of Participants with Medically Attended AEs (MAAEs), Serious AEs (SAEs), AEs of Special Interest (AESIs), and AEs Leading to Discontinuation | Day 1 up to Day 181 (End of study)
Geometric Mean Titer (GMT) of Serum RSV-A Neutralizing Antibodies (Abs) at Day 29 | Day 29
GMT of Serum RSV-B Neutralizing Abs at Day 29 | Day 29

SECONDARY OUTCOMES:
GMT of Serum RSV-A Neutralizing Abs | Day 1 up to Day 181 (End of study)
Geometric Mean Fold Rise (GMFR) of Serum RSV-A Neutralizing Abs | Day 181
GMT of Serum RSV-B Neutralizing Abs | Day 1 up to Day 181 (End of study)
GMFR of Serum RSV-B Neutralizing Abs | Day 181
Percentage of Participants With Seroresponse in RSV-A Neutralizing Abs | Day 181
Percentage of Participants With Seroresponse in RSV-B Neutralizing Abs | Day 181
Percentage of Participants With ≥2-fold Increase From Baseline in RSV-A Neutralizing Ab Titers | Day 181
Percentage of Participants With ≥2-fold Increase From Baseline in RSV-B Neutralizing Ab Titers | Day 181

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Velocity Clinical Research, Denver, Denver, Colorado
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research, Covington, Covington, Louisiana
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Velocity Clinical Research, Lincoln, Lincoln, Nebraska
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Velocity Clinical Research, Austin, Austin, Texas
  - Velocity Clinical Research, Hampton, Hampton, Virginia
  - Velocity Clinical Research, Spokane, Spokane, Washington